CLINICAL TRIAL: NCT04868461
Title: Effects of Protein Beverages Differing in Their Lubricating Properties on Appetite Control, Subsequent Food Intake and Salivary Biomarkers
Brief Title: Effect of Oral Lubrication on Appetite, Food Intake and Salivary Biomarkers in Protein Beverages
Acronym: LubSat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Anwesha Sarkar, Professor of Colloids and Surfaces, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LUBSAT (18-049) - Protein; 757993 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Appetitive Behavior
Keywords: Lubrication; protein; satiety; appetite control; food intake; salivary biomarkers
MeSH Terms: conditions — Appetitive Behavior | interventions — Beverages; Caseins; Crk-Associated Substrate Protein; Water

STUDY DESIGN:
Intervention Model Description: Tightly controlled cross-over study design with four arms.
Who Masked: Participant
Masking Description: This is a single-blind study i.e. participants do not know the real purpose of the study. They are given a cover story. They are told about the real purpose of the study at the completion of this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unheated whey protein (UWP) (Active Comparator): Participants are given a preload of 200 mL of unheated whey protein (UWP) in the morning, on a fasting state. After 30 minutes after the preload, participants are given ad libitum breakfast. They are asked to eat "as much or as little as they want, until they feel comfortably full".
  Interventions: Dietary Supplement: Unheated Whey Protein (UWP) beverage
- Heated whey protein (HWP) (Active Comparator): Participants are given a preload of 200 mL of heated whey protein (HWP) in the morning, on a fasting state. After 30 minutes after the preload, participants are given ad libitum breakfast. They are asked to eat "as much or as little as they want, until they feel comfortably full".
  Interventions: Dietary Supplement: Heated Whey Protein (HWP) beverage
- Casein (Cas) (Active Comparator): Participants are given a preload of 200 mL of Casein (Cas) in the morning, on a fasting state. After 30 minutes after the preload, participants are given ad libitum breakfast. They are asked to eat "as much or as little as they want, until they feel comfortably full".
  Interventions: Dietary Supplement: Casein (Cas) beverage
- Water (Placebo Comparator): The water has the same banana flavor and sweetness to match the protein beverages. Participants receive the same amount of water like protein beverages - 200mL.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Unheated Whey Protein (UWP) beverage — The preload is made from whey protein powder. The energy load of the preload is 119.7 kcal and has banana flavor and sweetener.
  Arms: Unheated whey protein (UWP)
Dietary Supplement: Heated Whey Protein (HWP) beverage — The preload is made from whey protein powder of 95% and it is heated for a certain amount of time. The energy load of the preload is 119.7 kcal and has banana flavor and sweetener.
  Arms: Heated whey protein (HWP)
Dietary Supplement: Casein (Cas) beverage — The preload is made from casein powder. The energy load of the preload is 105 kcal and has banana flavor and sweetener.
  Arms: Casein (Cas)
Dietary Supplement: Water — The preload is water acting as a control and contain the same banana flavor and sweetener to match the other three intervention - protein beverages.
  Arms: Water

SUMMARY:
The main aim of this study is to elucidate the influence of protein beverages differing in their lubrication properties (low/medium/high lubricating) and control (water) on satiety and satiation.

DETAILED DESCRIPTION:
The researchers propose an acute, randomized cross-over study that compares three types of protein beverages differing in their lubricating properties, i.e. one with low lubricating properties made using sodium caseinate, one with medium lubricating properties made by whey protein, and the third one with high lubricating properties made by heated whey protein. All three beverages contain added banana flavour and non-nutritive sweetener. Water acts as a control and has the same flavour and sweetness to match those of the protein beverages.

Participants are asked to come to the laboratory on four occasions. Before participating, each participant is screened for eligibility criteria using an online health screening questionnaire and Three Factors Eating Questionnaire. Participants are offered one of the four treatments (water or either of the three protein beverages), the order of which is randomized and counterbalanced.

Participants are instructed to fast for 11 hours and to restrict from drinking alcohol for 24 hours before each session. Each session lasts 1.5 hours (8.40 am until 10.10 pm). In the first session, weight and height are measured. Participants then provide baseline (- 5 min) appetite ratings on a 100 mm visual analogue scale (VAS). After that they are given the preload - either protein beverages differing in their lubricating properties or water. Then, participants are asked to rate their appetite on a 100-mm VAS every 10 minutes for the next 30 minutes. Ad libitum food is offered as breakfast after 30 min after ingesting the preload and the last VAS is taken. Saliva is taken three times during each session before preload, after preload consumption and before ad libitum breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years old
* With a BMI between 18.5 - 27.99 kg/m²)
* Generally healthy

Exclusion Criteria:

* have any blood borne disease;
* have type-1 or type-2 diabetes;
* have liver and kidney disease;
* have past history of gastrointestinal surgery;
* are a smoker;
* have oral infections/ diseases;
* have chronic or acute health condition that may affect ability to sense, eat, digest, absorb or excrete food;
* have a sensitive stomach (Irritable Bowel Stomach);
* are currently using prescribed or non-prescribed medication;
* are pregnant or lactating;
* are suffering from an illness, feeling unwell, having fever, or cold or cough;
* history of food allergy or intolerance;
* are on any special diet or are taking protein and/or fibre supplements;
* cannot tolerate protein beverages;
* present any COVID related symptoms (high temperature, a new continuous cough, a loss or change to your smell or taste);
* if you are self-isolating or if you leave with someone self-isolating or presenting COVID related symptoms.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Baseline level and change in hunger ratings | -5 minutes, 0 minute, 10 minutes, 20 minutes, 30 minutes, 50 minutes.
  A questionnaire assessing perceived hunger is completed at specific times points throughout each of the 1.5-h testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How hungry do you feel right now?" with anchors of "not all" to "extremely." The range is 0 mm (min hunger) and 100 is (max hunger).
Baseline level and change in fullness ratings | -5 minutes, 0 minute, 10 minutes, 20 minutes, 30 minutes, 50 minutes.
  A questionnaire assessing perceived fullness is completed at specific times points throughout each of the 1.5-h testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How full do you feel right now?" with anchors of "not all" to "extremely." The range is 0 mm (min fullness) and 100 is (max fullness).
Baseline level and change in desire to eat ratings | -5 minutes, 0 minute, 10 minutes, 20 minutes, 30 minutes, 50 minutes.
  A questionnaire assessing perceived desire to eat is completed at specific times points throughout each of the 1.5-h testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How strong is your desire to eat right now?" with anchors of "not all" to "extremely." The range is 0 mm (min desire to eat) and 100 is (max desire to eat).
Baseline level and change in prospective food consumption ratings | -5 minutes, 0 minute, 10 minutes, 20 minutes, 30 minutes, 50 minutes.
  A questionnaire assessing perceived prospective food consumption is completed at specific time points throughout each of the 1.5-h testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How much food do you think you could eat right now?" with anchors of "not all" to "extremely." The range is 0 mm (min prospective food consumption) and 100 is (max prospective food consumption.
Baseline level and change in thirst ratings | -5 minutes, 0 minute, 10 minutes, 20 minutes, 30 minutes, 50 minutes.
  A questionnaire assessing perceived thirst is completed at specific time points throughout each of the 1.5-h testing days. The questionnaire is a 100 mm VAS representing a horizontal line rating scale for each response. It asks: "How thirsty do you feel right now?" with anchors of "not all" to "extremely." The range is 0 mm (min thirst) and 100 is (max thirst).
Baseline level and change in breakfast energy intake | -5 minutes, 0 minute, 10 minutes, 20 minutes, 30 minutes, 50 minutes.
  The participants are provided with an ad libitum breakfast of cereals and milk, tea/coffee (at participant choice) and water. The amount of breakfast is provided (in grams) and is weighted prior to consumption and any remains are re-weighted after consumption. Energy consumed will be calculated. Participants are given 15 minutes for consuming the breakfast.
Baseline level and change in salivary protein | -5 minutes, 20 minutes, 50 minutes
  Saliva is collected on three time points on each visit. Salivary protein will be analyzed to determine the relationship between these components that affect oral lubrication and satiety and satiation.
Baseline level and change in salivary amylase | -5 minutes, 20 minutes, 50 minutes
  Saliva is collected on three time points on each visit. Salivary amylase will be analyzed to determine the relationship between these components that affect oral lubrication and satiety and satiation.
Baseline level and change in salivary mucin | -5 minutes, 20 minutes, 50 minutes,
  Saliva is collected on three time points on each visit. Salivary mucin will be analyzed to determine the relationship between these components that affect oral lubrication and satiety and satiation.

SECONDARY OUTCOMES:
Liking and wanting of the preload using Visual Analogue Scale (VAS) | Immediately after eating the preload.
  Liking and wanting of both the protein beverages and water are assessed through a 100 mm VAS scale where 0 means "not at all" and 100 means "extremely". Within the liking the ratings are taking on following attributes: the texture, flavor, sweetness and overall liking/pleasantness. The questions asked are: "How much did you like the texture of the product you have just consumed?", "How much did you like the flavor of the product you have just consumed?", How intense was the sweet taste of the product you have just consumed?", "How pleasant was the product you have just consumed? "with anchors from "not at all" to "extremely". And for the wanting assessment the question is: "How much did you want to consume the product you have just had?" with anchors from "not at all" to "extremely".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No